CLINICAL TRIAL: NCT03555110
Title: Effects of EMDR Therapy in Patients With Severe Obesity Submitted to Bariatric Surgery
Brief Title: Effects of EMDR Therapy in Patients With Severe Obesity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Roberto de Cleva, Principal Investigator, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 78695317.3.0000.0068
Record Dates: First submitted 2018-05-09; First posted 2018-06-13 (Actual); Last update posted 2019-10-10 (Actual); Status verified 2019-10

CONDITIONS: Obesity; Emotional Trauma
Keywords: EMDR Therapy; Bariatric Surgery; Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Controlled Group (Active Comparator): 30 morbid obese patients, 30 to 55 years old, submitted to Personality Factor Battery Test (PFB Test) during the study with the same frequency and criteria of the group of EMDR .
  Interventions: Behavioral: Personality Factor Battery Test (PFB Test)
- EMDR Group (Active Comparator): 30 morbid obese patients, 30 to 55 years old, submitted to Eye Movement Desensitization and Reprocessing Therapy (EMDR) during the study with the frequency of Twelve sessions, including:
  * Three evaluation and preparation sessions,
  * Eight EMDR sessions weekly with variable length of 60 minutes and
  * One closing session. The total intervention time will be about 3 (three) months. After the end of the 12 sessions of EMDR therapy, the patient will be evaluated again individually to verify the existence of change in PFB test results about the 5 big factors. The instrument will also be reapplied three months, twelve months and thirty-six months after bariatric surgery.
  Interventions: Behavioral: Eye Movement Desensitization and Reprocessing Therapy (EMDR)

INTERVENTIONS:
Behavioral: Personality Factor Battery Test (PFB Test) — Psychological instrument built for personality evaluation from the model of the Five Great Factors (FGF), that includes the following dimensions: Neuroticism, Extroversion, Socialization, Effort / Commitment), focusing on the component of the aspects of Neuroticism.
  Arms: Controlled Group
Behavioral: Eye Movement Desensitization and Reprocessing Therapy (EMDR) — It is a psychotherapeutic approach effective on treatment for trauma and post-traumatic stress disorder. It is an intervention that allows the desensitization of negative emotions from traumatic experiences.This therapy modifies memories that have been processed non-adaptively and become painful and dysfunctional memories. During the procedure, the patient is encouraged to move the eyes from side to side, associating these movements with a "target" situation, previously defined at the beginning of the session. The ocular movements can be replaced by tactile or sonorous stimuli. The series of stimuli must continue until the memory of the traumatic event can be reprocessed adaptively, that is, without the emotional, negative or painful process associated with that memory.
  Arms: EMDR Group

SUMMARY:
The aims of the study are to perform psychological intervention using EMDR Therapy (Eye Movement Desensitization and Reprocessing Therapy) in the preoperative period, evaluate the personality of each patient through the PFB test (Personality Factor Battery Test) at different times, compare the results obtained in the PFB test at different times of application and verify the existence of changes in the five major Personality Factors: Neuroticism, Extroversion, Socialization, Realization and Openness.

DETAILED DESCRIPTION:
Obesity is a multi-factorial disease requiring a multi-professional approach. Psychological causes also contribute to the development and maintenance of obesity. Traumatic experiences may be a risk factor for it as well. Emotional issues of obese patient often interfere with the results of bariatric surgery, where a large number of bariatric patients regain the weight or change symptoms.

The aim of the Effects of EMDR therapy with Severe Obesity Bariatric Surgery Patients randomized controlled trial is to determine the effects of 11 sessions of EMDR therapy, prior to surgery as compared to a control group. The Big Five personality factors will be used to evaluate the results. Both groups of patients will complete the Factorial Personality Battery, before the surgery, and 6 months and 12 months following bariatric surgery.

The initial hypothesis is that EMDR therapy will provide sufficient changes after surgery in the personality dynamics of obese patients, which will in turn favor emotional balance and weight maintenance as compared to the control group.

ELIGIBILITY:
Inclusion Criteria:

* both sexes
* BMI between 40 Kg/m2 and 50 Kg/m2
* ages between 30 and 55 years,
* minimum level of Elementary School, previously evaluated psychologically by the Psychology Service - University of São Paulo Medical School

Exclusion Criteria:

* history of severe personality disorders: psychotic symptoms or schizophrenia; bipolar disorder or dementia - groups A and B (DSM - IV);
* patients who present severe dissociative disorders (score above 25%), evaluated through the Dissociative Experiences Scale (DES);
* patients with heart problems and current pregnancy, with information obtained through the participants' reports.

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-06-02 (Actual); Study Completion 2020-06-02 (Estimated)

PRIMARY OUTCOMES:
change in emotional balance | Postoperative (3 months, 12 months and 36 months after bariatric surgery)
  This will be evaluated by the Factorial Personality Battery before and after surgery

SECONDARY OUTCOMES:
Total Weight loss | Postoperative (3 months, 12 months and 36 months after bariatric surgery)
  weight loss measured in percentage of weight loss (%WL)

CONTACTS AND LOCATIONS:
Overall Officials: Roberto De Cleva, Principal Investigator — Hospital das Clinicas da Faculdade de Medicina da USP
Locations (1):
- Hospital das Clinicas da Faculdade de Medicina da USP, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
The plan is to publish the complete data after the end of the study

REFERENCES:
- [Background] Alvarez J, Pavao J, Baumrind N, Kimerling R. The relationship between child abuse and adult obesity among california women. Am J Prev Med. 2007 Jul;33(1):28-33. doi: 10.1016/j.amepre.2007.02.036. PMID 17572308
- [Background] Cordas TA, Lopes Filho AP, Segal A. [Eating disorder and bariatric surgery: a case report]. Arq Bras Endocrinol Metabol. 2004 Aug;48(4):564-71. doi: 10.1590/s0004-27302004000400019. Epub 2005 Mar 7. Portuguese. PMID 15761522
- [Background] Felitti VJ, Anda RF, Nordenberg D, Williamson DF, Spitz AM, Edwards V, Koss MP, Marks JS. Relationship of childhood abuse and household dysfunction to many of the leading causes of death in adults. The Adverse Childhood Experiences (ACE) Study. Am J Prev Med. 1998 May;14(4):245-58. doi: 10.1016/s0749-3797(98)00017-8. PMID 9635069
- [Background] Perkonigg A, Owashi T, Stein MB, Kirschbaum C, Wittchen H-U. Posttraumatic stress disorder and obesity: evidence for a risk association. Am J Prev Med. 2009 Jan;36(1):1-8. doi: 10.1016/j.amepre.2008.09.026. Epub 2008 Oct 31. PMID 18976880
- [Background] Shapiro, F. Dessensibilização e Reprocessamento Através de Movimentos Oculares: Princípios Básicos, Protocolos e Procedimentos. (2a. ed.) - Brasília: Nova Temática, 2007